CLINICAL TRIAL: NCT06898580
Title: The Effect of Sacral Massage With a Tennis Ball on Labor Pain and Comfort During the Intrapartum Period
Brief Title: Sacral Massage With a Tennis Ball on Labor Pain and Comfort During the Intrapartum Period
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, emine algül, Master Student, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IUC-EBE-EA-01
Record Dates: First submitted 2025-03-12; First posted 2025-03-27 (Actual); Last update posted 2025-05-13 (Actual); Status verified 2025-03

CONDITIONS: Pain Management; Birth Comfort; Massage Effect; Labor Pain
Keywords: sacral massage; pain management; tennis ball; comfort of birth; reducing pain; labor pain
MeSH Terms: conditions — Agnosia; Labor Pain

STUDY DESIGN:
Intervention Model Description: Two groups with a experimental and control
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- sacral massage with a tennis ball (Active Comparator): When the cervical dilatation in labor is 5-6 cm, 7-8 cm and 9-10 cm, the woman will be asked to mark the intensity of the pain she feels on the VAS scale before starting the procedure. Then, the researcher explains sacral massage to the pregnant woman. While performing this application, the researcher will apply pressure to the sacral area with a tennis ball in a circular motion so that the patient can feel but not feel pain. The application will be applied to the pregnant woman for a total of 3 contractions. 30 minutes after each procedure, the woman will be asked again to mark the intensity of the pain she feels on the VAS scale and to mark the Birth Comfort Scale.
  Interventions: Other: sacral massage with tennis ball
- control groups (No Intervention): Pregnant women in the control group will not undergo any intervention other than routine hospital practices.

INTERVENTIONS:
Other: sacral massage with tennis ball — When the cervical dilatation in labor is 5-6 cm, 7-8 cm and 9-10 cm, the woman will be asked to mark the intensity of the pain she feels on the VAS scale before starting the procedure. Then, the researcher explains sacral massage to the pregnant woman. While performing this application, the researcher will apply pressure to the sacral area with a tennis ball in a circular motion so that the patient can feel but not feel pain. The application will be applied to the pregnant woman for a total of 3 contractions. 30 minutes after each procedure, the woman will be asked to mark the intensity of the pain she feels on the VAS scale and mark the Birth Comfort Scale. The research will end when a total of 70 experimental groups and 70 control groups are reached.
  Arms: sacral massage with a tennis ball

SUMMARY:
Although pregnancy and labor are physiological events, the pain caused by uterine contractions during labor is among the most severe pains. This causes many women to fear labor. For this reason, control of labor pain should be one of the main goals of the care given to women in labor. Therefore, this study was designed to determine the effect of sacral massage with a tennis ball on labor pain and labor comfort in the intrapartum period.

DETAILED DESCRIPTION:
Pregnant women hospitalized in the maternity unit will be evaluated for compliance with the inclusion criteria. Women who meet the inclusion criteria and are willing to participate in the study will be randomized according to the simple random numbers table and the study group will be determined by the researcher by drawing lots. The purpose and stages of the study will be explained verbally to the women whose group is determined and the women will be asked to read and sign the Informed Voluntary Consent Form. Then, the Pregnancy Identification Form will be filled in by the researchers using the face-to-face interview method. Then the massage will be explained to the pregnant women in the experimental group and they will be asked to evaluate the Visual Analog Scale (VAS) before the procedure. While performing this application, the researcher will apply pressure to the sacral region with a tennis ball in a circular motion in a way that the patient can feel but not feel pain. The application will be applied to the pregnant woman for a total of 3 contractions. 30 minutes after each procedure, the woman will be asked to mark the intensity of the pain she feels on the VAS scale and to mark the Birth Comfort Scale.

ELIGIBILITY:
Inclusion Criteria:

* To be able to read and write Turkish,
* Being over 18 years old
* Being primiparous
* Singular foetus and head presentation
* Pregnancy at term (37-42 weeks)
* Those without risk factors during pregnancy
* Being in the active phase of labour in stage 1
* Women without any chronic diseases
* Those without a diagnosed psychiatric illness
* To agree to participate in the research

Exclusion Criteria:

* If the participant wishes to leave the study voluntarily
* Administration of any analgesic medication to reduce pain during labour
* Development of any of the unexpected maternal-fetal risk conditions during labour
* Having a caesarean section for any reason
* The pregnant woman has spine and bone structure problems.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — pregnant women
Enrollment: 140 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Labor pain | Cervical dilatation will assses from 5-6 cm, 7-8 cm and 9-10 cm until delivery.
  Visual Analog Scale (VAS) is a scale to measure pain and other subjective symptoms. It was as first introduced by Hayes and Patterson in 1921. The Scale maximum point is 10 and minimum point is zero. And as the scale score increases, the pain measure also increases.When cervical dilatation is 5-6 cm, the pregnant woman is asked to mark her pain score on a VAS (Visual Analog Scale) score from one to ten, and then massage is applied. After 30 minutes of massage, the pregnant woman is asked to rate the pain score on the VAS (Visual Analog Scale).

SECONDARY OUTCOMES:
birth comfort | Cervical dilatation will assses from 5-6 cm, 7-8 cm and 9-10 cm until delivery.
  Childbirth Comfort Questionnaire is a scale for assessing childbirth comfort. The validity and reliability of the scale was made by Potur et al. in 2014. The Scale maximum point is 45 and minumum point is nine. And as the scale score increases, the comfort level also increases.
  When cervical dilatation is 5-6 cm, the pregnant woman is asked to check the appropriate options on the 9-item scale on the CCQ. We want this procedure to be done three times in total when the pregnant woman is 5-6 cm, 7-8 cm and 9-10 cm.

IPD SHARING:
Plan to Share IPD: No